CLINICAL TRIAL: NCT03825848
Title: The Influence of Shunting Left/Right Portal Vein Branch on Post-transjugular Intrahepatic Portosystemic Shunt Hepatic Encephalopathy: a Multicenter Randomized Controlled Trial
Brief Title: The Influence of Post-transjugular Intrahepatic Portosystemic Shunt Hepatic Encephalopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2018-292R
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Portal Hypertension; Hepatic Encephalopathy
MeSH Terms: conditions — Hypertension, Portal; Hepatic Encephalopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Portal Vein Branch (Experimental): Shunt left portal vein branch during the trans jugular intrahepatic portal systemic shunt
  Interventions: Procedure: trans jugular intrahepatic portal systemic shunt
- Right Portal Vein Branch (Experimental): Shunt right portal vein branch during the trans jugular intrahepatic portal systemic shunt
  Interventions: Procedure: trans jugular intrahepatic portal systemic shunt

INTERVENTIONS:
Procedure: trans jugular intrahepatic portal systemic shunt — Shunting left or right PV branch in the TIPS procedure

SUMMARY:
Through a multicenter randomized controlled trial of TIPS to prevent post-hepatitis B cirrhosis of esophagogastric varices, the incidence of hepatic encephalopathy, the rate of stent patency, the incidence of rebleeding and survival in the left and right branches of the portal vein were compared.

DETAILED DESCRIPTION:
The most common cause of cirrhosis in China is hepatitis B virus infection; post-hepatitis B cirrhosis with gastroesophageal variceal hemorrhage is common in clinical practice; recent studies [14] found that implantation of 8 mm diameter is compared with the use of 10 mm diameter stents. The membrane stent significantly reduced the incidence of HE after TIPS without affecting the shunt effect. To further evaluate the effect of "left/right branch of shunt portal" on hepatic encephalopathy after TIPS, we intend to conduct the following studies: for individual etiology (post-hepatitis B cirrhosis), the only indication (to prevent recurrent rupture of gastroesophageal varices) ), implanted 8mm diameter Viatorr stent, unified HE evaluation criteria, and stratified multi-center randomized clinical trial study with Child classification, hope to guide TIPS in line with China's national conditions through the high-level evidence-based medical evidence obtained.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's gender is not limited, ≥ 18 years old and ≤ 75 years old;
2. Clinically diagnosed post-hepatitis B cirrhosis;
3. History of esophageal varices venous rupture confirmed by endoscopy, re-bleeding after standard treatment;
4. Liver function Child A or B;
5. Imaging (CT or MRI) suggests that the left/right first branch of the intrahepatic portal can construct a shunt;
6. Platelet count ≥ 50 × 109 / L;
7. Prothrombin time (PT) does not exceed the upper limit of the normal control for 3 seconds;
8. Serum creatinine concentration ≤115umol/L;
9. Patients and their families agree to join the clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Imaging confirms portal vein thrombosis;
2. Patients who have undergone previous surgical treatment of portal hypertension (including splenectomy, surgical disconnection or shunt);
3. Combine any malignant tumor;
4. History of previous hepatic encephalopathy;
5. Consolidation of intractable ascites;
6. Pulmonary artery pressure > 40 mmHg, left ventricular ejection fraction < 50%, congestive heart failure or severe valvular insufficiency;
7. Others: persistent active bleeding, vital signs can not be maintained, blood ammonia ≥ 100, total bilirubin > 51umol / L failed to improve after symptomatic treatment; combined active infection, especially biliary system inflammation; female patients are pregnant Or lactation; severe contrast allergy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of HE | 2 years
  compare difference incidence of HE between shunting left and right portal vein branch

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Luo, doctor, Study Chair — Fudan University
Locations (1):
- Department of Interventional Radiology, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wang Q, Lv Y, Bai M, Wang Z, Liu H, He C, Niu J, Guo W, Luo B, Yin Z, Bai W, Chen H, Wang E, Xia D, Li X, Yuan J, Han N, Cai H, Li T, Xie H, Xia J, Wang J, Zhang H, Wu K, Fan D, Han G. Eight millimetre covered TIPS does not compromise shunt function but reduces hepatic encephalopathy in preventing variceal rebleeding. J Hepatol. 2017 Sep;67(3):508-516. doi: 10.1016/j.jhep.2017.05.006. Epub 2017 May 12. PMID 28506905
- [Result] American Association for the Study of Liver Diseases; European Association for the Study of the Liver. Hepatic encephalopathy in chronic liver disease: 2014 practice guideline by the European Association for the Study of the Liver and the American Association for the Study of Liver Diseases. J Hepatol. 2014 Sep;61(3):642-59. doi: 10.1016/j.jhep.2014.05.042. Epub 2014 Jul 8. No abstract available. PMID 25015420
- [Result] Bajaj JS, Heuman DM, Sterling RK, Sanyal AJ, Siddiqui M, Matherly S, Luketic V, Stravitz RT, Fuchs M, Thacker LR, Gilles H, White MB, Unser A, Hovermale J, Gavis E, Noble NA, Wade JB. Validation of EncephalApp, Smartphone-Based Stroop Test, for the Diagnosis of Covert Hepatic Encephalopathy. Clin Gastroenterol Hepatol. 2015 Oct;13(10):1828-1835.e1. doi: 10.1016/j.cgh.2014.05.011. Epub 2014 May 17. PMID 24846278
- [Derived] Ma J, Luo J, Zhang W, Zhou Y, Zhang Z, Yang M, Zhuang Z, Ma L, Yu J, Zhou X, Yan Z. The influence of shunting left/right portal vein branch on post-TIPS hepatic encephalopathy: a study protocol for multicenter randomized blinded controlled trial. Trials. 2023 May 6;24(1):312. doi: 10.1186/s13063-023-07326-9. PMID 37149647